CLINICAL TRIAL: NCT00389545
Title: Intracoronary Stem Cells in Large Myocardial Infarction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charles University, Czech Republic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IGA 8225
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2006-10-19 (Estimated); Status verified 2006-10

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

INTERVENTIONS:
Procedure: Intracoronary infusion of autologous bone-marrow derived stem cells

SUMMARY:
Despite the widespread use of effective reperfusion therapies, the patients presenting late with large myocardial infarction have poor outcomes. The aim of the study was to investigate the safety and efficacy of intracoronary injection of autologous bone marrow-derived mononuclear cells (BMNCs) in patients with large myocardial infarction

DETAILED DESCRIPTION:
In the current era, up to 30% of patients with ST-segment elevation myocardial infarction, usually those presenting late, show ongoing left ventricular (LV) remodeling and poor clinical outcome despite primary percutaneous coronary intervention (PCI). Cardiac transfer of bone marrow-derived stem and progenitor cells has been investigated as an adjunctive therapy to promote regeneration of infarcted myocardium. Therefore, we designed a multicenter, randomized study to test the safety and efficacy of intracoronary injection of autologous BMNCs in patients with large acute anterior myocardial infarction and late presentation, who were treated with successful primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the first ST-segment elevation acute anterior myocardial infarction due to occlusion of the proximal left anterior ascending coronary artery (LAD), who will underwent successful primary stented PCI. Patients are eligible if they have primary PCI from 4 to 12 hours after symptoms onset and show reduced LV ejection fraction ≤ 45% with at least 3 akinetic segments in the LAD perfusion territory at echocardiogram performed 24 hours after PCI.

Exclusion Criteria:

* Exclusion criteria are age ≥ 80 years, cardiogenic shock (Killip IV), multivessel coronary artery disease, serious renal or hepatic disease, blood cells disorders, documented cancer or terminal illness.

Ages: 18 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Martin Penicka, Principal Investigator — Charles University, Prague, Czech Republic